CLINICAL TRIAL: NCT02434406
Title: Feasibility of a Web-Based Intervention for Women With Postpartum Anxiety: A Randomized Controlled Trial
Brief Title: Website-Based Self-Help for Women With Anxiety After Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PhD/14-15/16
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Anxiety Disorders
Keywords: Anxiety; Anxiety disorders; Mental health; Postpartum period; maternal welfare; internet; intervention studies; feasibility studies; randomized controlled trial; patient acceptance of health care
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based intervention (Experimental): Participants get access to the web-based intervention and are asked to work through the 8 modules of the intervention within eight weeks. The intervention program sends automated weekly email reminders about the current session. In addition, users are offered weekly optional 30-minute telephone support with a trained intervention coach.
  Interventions: Behavioral: internet-What Am I Worried About
- Wait-list control (No Intervention): Participants get standard care and will be offered access to the web-based intervention at 8-weeks post-randomization.

INTERVENTIONS:
Behavioral: internet-What Am I Worried About — This web-based intervention consists of three sections: 1) Is this for me? 2) Practice 3) Understanding. The three main sections are divided up into nine sessions. Participants will get access to the program for eight weeks and can access the sessions more than once. Sessions are made up of multimedia presentations and worksheets that are completed online.
  Arms: Web-based intervention

SUMMARY:
This study examines the feasibility and acceptability of a web-based intervention program for women with anxiety after childbirth, potential anxiety reduction after the intervention and determines the feasibility of the study design (randomized controlled design) and recruitment for the intervention in this population to inform the protocol (including effect size and study power) for a randomized controlled trial.

DETAILED DESCRIPTION:
Background: What Am I Worried About (WAWA) is a self-help booklet intervention for women experiencing anxiety after birth based on cognitive-behavioural and mindfulness principles developed in Australia. The WAWA booklet was found to be acceptable, safe, stigma free, feasible, and demonstrated preliminary efficacy in Australia. A web-based version of WAWA for the use in the United-Kingdom (UK) was developed at City University London in collaboration with the intervention development team in Australia. However, before dissemination the web-based version of WAWA (iWAWA) in the UK it is deemed important to evaluate the program. Therefore, this study aims to examine the feasibility, acceptability, and potential efficacy of this web-based intervention program for women with anxiety after childbirth in the UK.

The primary objectives of the proposed study are to:

conduct a randomized controlled trial and

* examine the feasibility of web-based treatment program (iWAWA) in terms of engagement and usability.
* examine user's acceptability of iWAWA in terms of usefulness, satisfaction, and credibility.

The secondary objectives of this study are to:

* obtain initial estimates of anxiety levels and examine potential patient improvement over the course of the intervention and compared to the control group.
* determine the feasibility of the study by examining recruitment, consent, attrition, follow-up rates, as well as response rates to questionnaires.

Method: For this feasibility study, an embedded mixed methods design is employed utilizing both quantitative and qualitative methods to achieve the above stated aims. For the quantitative part, a randomized control trial is conducted. Outcomes are assessed at pre-intervention, throughout the intervention, post-intervention, and 1-month post-intervention. For the qualitative part, semi-structured interviews are used for a more in-depth exploration of acceptability and feasibility of the iWAWA intervention. The interviews with participants are carried out post intervention.

Study benefits: Based on the participants' feedback, this study hopes to inform development and adaptation of the investigated web-based intervention. If the interventions acceptability and feasibility is confirmed, the next steps would be to test the intervention efficacy in a stage II randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* Women who are within the first 12 months postpartum (at the beginning of the intervention)
* Aged over 18
* Living in England
* Sufficient knowledge of written and spoken English
* Access to internet at home
* Report a score of ≥5 on the Generalized Anxiety Disorder Scale (GAD-7; Spitzer, Kroenke, Williams, & Löwe, 2006)

Exclusion Criteria:

* Still birth or perinatal death of latest baby
* Latest baby seriously ill
* Report self-harm or suicidal ideation
* Currently receiving formal psychotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-03-26 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Engagement as measured by the number of log-ins into the web-based intervention | At time of intervention (8 weeks)
Engagement as measured by the duration of log-ins into the web-based intervention | At time of intervention (8 weeks)
Engagement as measured by the total duration of time spent on the web-based intervention | At time of intervention (8 weeks)
Engagement as measured by the time spent on individual pages of the web-based intervention | At time of intervention (8 weeks)
Engagement as measured by the number of intervention coach calls | At time of intervention (8 weeks)
Usability as measured by participant's report of usefulness ("I found this module useful.") of each intervention module on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree). | At time of intervention (8 weeks) after each completed intervention module
Usability as measured by participant's report of clarity ("This module was clear and understandable.") of each intervention module on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree). | At time of intervention (8 weeks) after each completed intervention module
Usability as measured by participant's report of usability on the System Usability Scale (SUS) | Within 2 weeks after the intervention
  The System Usability Scale (SUS) is a 10-item instrument rated on 5-point Likert scale (1 = strongly disagree to 5 = strongly agree) and participants are asked to rate the degree to which they agree with positive and negative descriptions of a program. The SUS will be adapted for this study by replacing 'the system/product' with 'iWAWA' for all items. Higher scores indicate better usability.
Usability as measured by participant's report of usability on a series of items designed to measure ease-of-use and unobtrusiveness on 7-point Likert scale (1 = strongly disagree to 7 = strongly agree) | Within 2 weeks after the intervention
Usability as measured by participant's report of any technical problems experienced with the intervention website | Within 2 weeks after the intervention
Usability as measured by participant's report of interest in future usage of the intervention | Within 2 weeks after the intervention
Usefulness as measured by participant's report of a series of items designed to measure perceived usefulness on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree). | Within 2 weeks after the intervention
Satisfaction as measured by participant's report of a series of items designed to measure perceived satisfaction on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree). | Within 2 weeks after the intervention
Satisfaction as measured by participant's report on the Client Satisfaction Questionnaire (CSQ-8) | Within 2 weeks after the intervention
  The Client Satisfaction Questionnaire (CSQ-8) will further be used and adapted to assess satisfaction. The CSQ-8 consists of eight items which are rated on 5-point Likert scale. The CSQ-8 will be adapted for this study by substituting 'service' with 'help" and "program" with "iWAWA" in all items.
Credibility as measured by participant's report on the first 4 items of Credibility/ Expectancy Questionnaire (CEQ) | Within 2 weeks after the intervention
  The Credibility/ Expectancy Questionnaire (CEQ) is a 6-item widely applied measure of the expectancies or perception of intervention credibility and will be adapted for the use in this study.
Women's perspectives and experiences as measured by semi-structured interviews | Within 8 weeks after the intervention
Engagement as measured by the duration of intervention coach calls | Continuous throughout the 8 week intervention period
Usability as measured by participant's report of hypothetical recommendation of the intervention to others. | Within 2 weeks after the intervention

SECONDARY OUTCOMES:
Anxiety level as measured by participant's report on the Generalized Anxiety Disorder Scale (GAD-7) | Within 1 week before the intervention
  The Generalized Anxiety Disorder Scale (GAD-7) is a seven-item anxiety measure and items are rated on 4-point Likert-scale ranging from 0' (not at all) to '3' (nearly every day).
Depression, anxiety and stress symptomatology as measured by participant's report on the Depression, Anxiety, and Stress Scale (DASS 21) | Within 1 week before the intervention
  The Depression, Anxiety, and Stress Scale (DASS 21) is a 21-item self-report measure of current depressive, anxiety, and stress symptoms. Low positive affect, reduced self-esteem and motivation, and a sense of hopelessness is assessed by seven depression items; fearfulness and physiological arousal is assessed by seven anxiety items, and tension, irritability and a low threshold to frustration are measured by seven stress items. Higher scores indicate more severe symptoms.
Anxiety level as measured by participant's report on the Generalized Anxiety Disorder Scale (GAD-7) | Within 1 week after the intervention
  The Generalized Anxiety Disorder Scale (GAD-7) is a seven-item anxiety measure and items are rated on 4-point Likert-scale ranging from 0' (not at all) to '3' (nearly every day).
Depression, anxiety and stress symptomatology as measured by participant's report on the Depression, Anxiety, and Stress Scale (DASS 21) | Within 1 week after the intervention
  The Depression, Anxiety, and Stress Scale (DASS 21) is a 21-item self-report measure of current depressive, anxiety, and stress symptoms. Low positive affect, reduced self-esteem and motivation, and a sense of hopelessness is assessed by seven depression items; fearfulness and physiological arousal is assessed by seven anxiety items, and tension, irritability and a low threshold to frustration are measured by seven stress items. Higher scores indicate more severe symptoms.
Anxiety level as measured by participant's report on the Generalized Anxiety Disorder Scale (GAD-7) | Within 1 week after the end of the 4 week post-intervention follow-up period
  The Generalized Anxiety Disorder Scale (GAD-7) is a seven-item anxiety measure and items are rated on 4-point Likert-scale ranging from 0' (not at all) to '3' (nearly every day).
Depression, anxiety and stress symptomatology as measured by participant's report on the Depression, Anxiety, and Stress Scale (DASS 21) | Within 1 week after the end of the 4 week post-intervention follow-up period
  The Depression, Anxiety, and Stress Scale (DASS 21) is a 21-item self-report measure of current depressive, anxiety, and stress symptoms. Low positive affect, reduced self-esteem and motivation, and a sense of hopelessness is assessed by seven depression items; fearfulness and physiological arousal is assessed by seven anxiety items, and tension, irritability and a low threshold to frustration are measured by seven stress items. Higher scores indicate more severe symptoms.
Study feasibility as measured by recruitment rate | Within 4 weeks of ending recruitment
Study feasibility as measured by eligibility rate | Within 4 weeks of ending recruitment
Study feasibility as measured by consent rate | Within 4 weeks of ending recruitment
Study feasibility as measured by retention rate | Within 4 weeks of ending data collection
Study feasibility as measured by pre-intervention data collection rate | Within 4 weeks of ending data collection
Study feasibility as measured by pre-intervention data collection completeness | Within 4 weeks of ending data collection
Study feasibility as measured by post-intervention data collection rate | Within 4 weeks of ending data collection
Study feasibility as measured by post-intervention data collection completeness | Within 4 weeks of ending data collection
Study feasibility as measured by 4 week post intervention follow-up data collection rate | Within 4 weeks of ending data collection
Study feasibility as measured by 4 week post intervention follow-up data collection completeness | Within 4 weeks of ending data collection

CONTACTS AND LOCATIONS:
Overall Officials: Miriam T Ashford, MS, cand.PhD, Principal Investigator — City, University of London; Susan Ayers, Professor, Principal Investigator — City, University of London
Locations (2):
- United Kingdom (2):
  - City, University of London, London, Greater London
  - City University of London, London

REFERENCES:
- [Background] Rowe HJ; Calcagni SC; Galgut S; Michelmore J; Fisher, JRW. Self-management of mild to moderate anxiety in women who have recently given birth: Development and acceptability of a theoretically sound complex intervention. International Journal of Mental Health Promotion 2014 Oct; 16(5): 308-319. doi:10.1080/14623730.2014.964050
- [Derived] Ashford MT, Olander EK, Rowe H, Fisher JR, Ayers S. Feasibility and Acceptability of a Web-Based Treatment with Telephone Support for Postpartum Women With Anxiety: Randomized Controlled Trial. JMIR Ment Health. 2018 Apr 20;5(2):e19. doi: 10.2196/mental.9106. PMID 29678804